CLINICAL TRIAL: NCT00356798
Title: The Phase-I Clinical Trial Protocol for the Pandemic Inactivated Influenza Vaccine
Brief Title: Randomized, Double Blinded, Placebo Control Clinical Trial of Pandemic Influenza Inactive Vaccine on Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-PanFlu-1001
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2007-11

CONDITIONS: Influenza
Keywords: pandemic; influenza; H5N1; vaccine
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: an inactivated whole virion H5N1 vaccine, adjuvanted

SUMMARY:
Based on pre-clinical trial data and principle of GCP, the objective of phase I clinical trial is to evaluate safety and immunogenicity of Pan-flu vaccine, an inactivated whole virion H5N1 vaccine with aluminium hydroxide adjuvant.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age from 18 to 60 years old;
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process;
* Able and willing to complete the informed consent process.

Exclusion Criteria:

* Woman who is breast-feeding or planning to become pregnant during the following 210 days of study participation;
* Persons who engage in the following occupations: culturist, slaughter, sale and forwarder of avian;
* Subject has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine, such as egg, egg protein, etc;
* Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain;
* Autoimmune disease or immunodeficiency;
* Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids;
* Diabetes mellitus (type I or II), with the exception of gestational diabetes;
* History of thyroidectomy or thyroid disease that required medication within the past 12 months;
* Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years;
* Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws;
* Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of study;
* Seizure disorder other than 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years;
* Asplenia, functional asplenia or any condition resulting in the absence or removal o the spleen;
* Guillain-Barre Syndrome (GBS);
* Abnormal result of laboratory test as below:

  * Biochemistry assaying: Alanine Aminotransferase /Serum Glutamate Pyruvate Transaminase (ALT), Total Bilirubine Tbil (TBIL), Direct Bilirubine Tbil (DBIL), Blood Urea Nitrogen (BUN) and Creatinine (Cr).
  * Routine blood assaying, routine urine assaying.
  * HBsAg positive;
* Pregnancy test positive for female;
* Subject has received any of the following substances:

  * Immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis).
  * Blood products within 3 months prior to initial study vaccine administration.
  * Other study drug within 30 days prior to initial study vaccine administration. Live attenuated vaccines within 30 days prior to initial study vaccine administration.
  * Medically indicated subunit or killed vaccines, e.g. pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration.
  * Current anti-TB prophylaxis or therapy.
* Fever before vaccination, axillary temperature 37.0 centigrades.
* Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to enrollment.
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120
Dates: Start 2005-12; Study Completion 2006-04

PRIMARY OUTCOMES:
To evaluate the safety of pandemic inactivated influenza vaccine by different does.

SECONDARY OUTCOMES:
To evaluate the immunogenicity of pandemic inactivated influenza vaccine by different does.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangtao Lin, MD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Lin J, Zhang J, Dong X, Fang H, Chen J, Su N, Gao Q, Zhang Z, Liu Y, Wang Z, Yang M, Sun R, Li C, Lin S, Ji M, Liu Y, Wang X, Wood J, Feng Z, Wang Y, Yin W. Safety and immunogenicity of an inactivated adjuvanted whole-virion influenza A (H5N1) vaccine: a phase I randomised controlled trial. Lancet. 2006 Sep 16;368(9540):991-7. doi: 10.1016/S0140-6736(06)69294-5. PMID 16980114